CLINICAL TRIAL: NCT01090674
Title: Relationship Between Respiratory Functional Tests and Image Thoracic Techniques in Patients With Neuromuscular Diseases.
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: PR01/01/2007
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Diaphragmatic force; mobility
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with amyotrophic lateral sclerosis.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — We perform in all patients respiratory functional tests, thoracic x-ray, SNIF test and diaphragmatic magnetic resonance imaging.

SUMMARY:
It is very important monitoring respiratory muscle function in patients with amyotrophic lateral sclerosis (ALS). We have at our disposal Respiratory Functional Tests (forced vital capacity (FVC), maximal mouth-inspiratory force (MIF), maximal mouth-expiratory force (MEF), Cough Peak expiratory flow (cPEF), maximal voluntary ventilation (MVV), arterial blood gases and nocturnal pulsioxymetry) and Thoracic Image Techniques (inspiratory/expiratory Thorax x-ray and x-ray scope). But all this explorations present some technique limitations. They are two new methods to explore diaphragmatic function: SNIF test and Diaphragm magnetic resonance imaging (dMRI). SNIF test is simple and easy to be done and it can avoid some problems that have the other respiratory functional test in this kind of patients. dMRI seems to correlate with respiratory functional test and it can be useful monitoring diaphragmatic mobility. The objective of our study is to compare and to correlate SNIF test and dMRI with x-ray techniques and respiratory functional tests that measure diaphragmatic force and function. First of all we will study 10 healthy people with a forced spirometry, MIF, MEF and dMRI, trying to obtain diaphragmatic mobility reference values with dMRI. Lately, we will study patients with ALS. In the first place, we will perform a transversal study with 30 patients. We will do a forced spirometry, MIF, MEF, MVV, cPEF, SNIF, arterial blood gases and nocturnal pulsioxymetry, forced Inspiratory and expiratory Thorax x-ray, diaphragmatic x-ray scope and dMRI. Secondly, we will perform a prospective study, where we will analyze these variables evolution at 3 and 6 months. We hope we can apply the two new techniques in the future because we think they are simpler, more accurate and more objective to evaluate diaphragmatic mobility.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic lateral sclerosis patients.
* Clinically stable, at least for one month.

Exclusion Criteria:

* Claustrophobic patients.
* Patients using continuous non-invasive ventilation treatment.
* Incapacity to tolerate supine decubitus.
* Incapacity to execute respiratory functional tests.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with amyotrophic lateral sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2007-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Different measures of diaphragmatic mobility, force and function. | One year
  To compare and correlate all different image techniques that evaluate diaphragmatic mobility with all different respiratory functional variables that measure diaphragmatic (and muscular in general) force and function.

SECONDARY OUTCOMES:
Diaphragmatic MRI usefulness | One year
  * To evaluate dMRI usefulness in monitoring diaphragmatic mobility.
  * To evaluate if we can establish a value of diaphragm mobility (in mm) observed with dMRI to suggest the initiation of non invasive ventilation treatment.
  * To evaluate if dMRI can predict ALS prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain